CLINICAL TRIAL: NCT00837408
Title: Genetics of Type 2 Diabetes Among Han Chinese
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999909071; 09-HG-N071
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Diabetes; Hypertension
Keywords: GWAS
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Individuals with Type 2 Diabetes
- Controls: Individuals without Type 2 Diabetes

SUMMARY:
Objectives:

* To conduct a genome-wide association study (GWAS) to identify susceptibility genetic variants for diabetes among Han Chinese.
* To conduct resequencing of positional candidate gene/loci to identify likely functional variants in a subset of the cohort.
* To conduct replication studies of the top-100 scoring variants in three independent African and European ancestry samples.
* To investigate whether diabetes-associated variants discovered in European populations increase diabetes risk in Han Chinese.

Eligibility:

* Patients 25 years of age with newly diagnosed T2D in Suizhou, China. Control subjects are nondiabetics, age and ethnically matched to patients.

Design:

* The study design for both patients and controls consists of the following steps:
* Discuss informed consent process and obtain signed informed consent form. Informed consent will be administered by trained clinic staff.
* Assign study ID (barcode)
* Administer questionnaires
* Obtain spot urine sample
* Measure blood pressure
* Obtain anthropometric measurements including body composition
* Perform finger prick for blood glucose level
* Obtain venous blood samples
* Perform eye examination
* On the following day, perform confirmatory blood glucose for the small subset of participants requiring confirmation of previous test result
* DNA extraction of stored samples will be done at either the National Institutes of Health or the laboratory in China.
* GWAS will be conducted using publicly available software packages.

DETAILED DESCRIPTION:
This research protocol is designed to study the genetic basis of Type 2 Diabetes (T2D) in Han Chinese. This project taking place at Suizhou Central Hospital complements several years of similar research activities conducted by Dr. Rotimi s lab in populations of the African Diaspora with study sites in Nigeria, Ghana, Kenya and the US. Suizhou Hospital was selected because of the existence of an excellent team of research investigators, infrastructure and more importantly, the availability of a large population from which to enroll and examine persons with diabetes and normal controls. Previous funding from Dr. Rotimi s lab at Howard University made it possible for Dr. Jiang and staff to enroll 1000 cases and controls. Therefore, the goal of the current project is to enroll additional 1500 cases of T2D and 1500 ethnically matched Han controls from Suizhou to facilitate the conduct of genome-wide association study (GWAS) and candidate gene/loci studies in Han, Chinese. The current project will increase the number of subjects for future GWAS, linkage disequilibrium (LD) mapping and functional studies to over 4,000 ethnically balanced cases (greater than 2,000) and controls (greater than 2,000). Identified candidate genes/loci will be investigated by re-sequencing and functional studies will be conducted to identify susceptibility variants for diabetes and associated complications including obesity, hypertension, nephropathy, neuropathy and retinopathy. Given past activities, it is also anticipated that this resource will form the basis of multiple collaborations between Dr. Rotimi s lab, several NIH intramural researchers and non-NIH scientists.

ELIGIBILITY:
* INCLUSION CRITERIA:

Cases Men and women with confirmed type 2 diabetes mellitus that are either on treatment for diabetes or newly diagnose with blood sugar reading on more than one occasion exceeding or equal to 126 mg/dl. These persons must be above the age of 25 years. In this regard, all newly diagnosed participants will be required to visit the clinic on the following day to perform fasting blood glucose test to confirm previous results.

Controls Men and women with fasting plasma glucose (FPG) less than 100 mg/dl (5.6 mmol/l). Controls must be above age 25 years and should be ethnically matched to the cases. Enrolled cases and controls have to be unrelated. Therefore, only one person may be enrolled from each family unless they are husband and wife.

Attempts will be made to enroll an equal number of men and women. To ensure that ethnic distribution is maintained in the parent study, we are proposing to enroll only Han Chinese participants.

EXCLUSION CRITERIA:

People who do not meet the above criteria (e.g., younger than 24, without the blood sugar requirements, etc). No more than one non-spouse member of each family. No prisoners, pregnant women or fetuses will be included in this study.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases will be drawn from Type 2 Diabetics attending clinics at the Suizhou Central Hospital. Controls will be ethnicity-matched individuals from the community served by this hospital.
Sampling Method: Non-Probability Sample
Enrollment: 2379 (Actual)
Dates: Start 2009-02-03 (Actual); Primary Completion 2012-02-03 (Actual); Study Completion 2012-02-03 (Actual)

PRIMARY OUTCOMES:
Type 2 Diabetes | Cross-sectional
  Diagnosis of type 2 diabetes based on blood glucose measurement.

CONTACTS AND LOCATIONS:
Overall Officials: Charles N Rotimi, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- HuBei Suizhou Central Hospital, Suizhou, China